CLINICAL TRIAL: NCT00671450
Title: Visual Dysfunction in MTBI: A Comparison Group Study
Brief Title: Visual Dysfunction in Mild Traumatic Brain Injury (MTBI): A Comparison Group Study
Acronym: VDMTBI
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: SHP 08-142
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2009-08

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Participants will be patients diagnosed with PTSD but with no history of TBI. Participants must be between the ages of 19 and 39. Participants must be compentent to sign a consent form and be willing ot participate in a vision screening.

SUMMARY:
In an on-going study of visual characteristics of personnel diagnosed with a mild traumatic brain injury (MTBI) related to their service in Iraq and Afghanistan we found a high rate of binocular vision problems (such as double/blurry vision, reading difficult, etc.). These individuals are also usually diagnosed with post traumatic stress disorder (PTSD). PTSD is known to cause some vision symptoms. We wish to conduct this study on individuals with PTSD (but not an MTBI) to see if they have symptoms similar to those in individuals who have MTBI. This will provide us with information useful in determining the specific cause of the visual symptoms in the MTBI population.

DETAILED DESCRIPTION:
We will recruit 75 patients diagnosed with PTSD, but with no history of mild traumatic brain injury (MTBI), from the population of the VAPAHCS PTSD Center and Clinics. These volunteers will be scheduled for an eye screening developed for a concurrent project to assess visual dysfunction (accommodation/vergence insufficiency, pursuit/saccade deficits, etc.) in patients diagnosed with MTBI and seen at the Palo Alto Polytrauma Network Site clinic. The MTBI patients have unexpectedly high rates of binocular dysfunction, although their visual acuities and visual fields are normal/near normal. The MTBI diagnosis is associated with a combat blast event in some 90% of cases. Th majority of this population has also been diagnosed with PTSD. PTSD is known to cause some visual symptoms, thus it is necessary for us to determine if the visual dysfunctions in the MTBI are related to their PTSD diagnosis or not. The volunteer participants will be scheduled for an eye screening and consented prior to the screening. Inclusion criteria include diagnosis of PTSD, aged 19 to 39, and willingness to participate. Exclusion criteria is primarily history of TBI. The visual screen includes assessments of visual acuity, visual field, self-reported visual function (i.e., light sensitivity, eye fatigue, reading difficulty), and measures of accommodative function, vergence, pursuit and saccades. The data collected will be compared to the data from the ongoing study of visual dysfunction in patients diagnosed with MTBI.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PTSD
* no history of MTBI
* between 19 and 39 years of age
* a veteran

Exclusion Criteria:

* a history of MTBI
* over the age of 39
* an unwillingness to participate

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be drawn from the patient population of the VAPAHCS PTSD Center and Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Presence or absence of binocular dysfunction | The primary outcome will be measured at a single visual screen lasting approximately one hour.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Goodrich, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States